CLINICAL TRIAL: NCT06227975
Title: A Phase 1, Single-center, Open-label Study to Evaluate the Absorption, Metabolism, and Excretion of Orally Administered [14C]-BMS-986368 in Healthy Male Participants
Brief Title: A Study to Evaluate the Absorption, Metabolism, and Excretion of Orally Administered [14C]-BMS-986368 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM045-1003
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers
Keywords: ADME; Healthy male volunteers; Pharmacokinetics; BMS-986368; CC-97489

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-BMS-986368 (Experimental)
  Interventions: Drug: [14C]-BMS-986368

INTERVENTIONS:
Drug: [14C]-BMS-986368 — Specified dose on specified days
  Other Names: CC-97489

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics (PK), metabolites, route of elimination, and mass balance of BMS-986368 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants as determined by no clinically significant deviations from normal in medical history, physical examination, vital signs, 12-lead ECGs, and clinical laboratory determinations, as assessed by the investigator.
* Body mass index of 18.0 to 35.0 kg/m2, inclusive. Body mass index = weight (kg)/(height[m])^2

Exclusion Criteria:

* History of hypokalemia.
* Any significant acute or chronic medical illness as determined by the investigator.
* Participant has a history of syncope in the year prior to Day 1.

Other protocol-defined incusion/exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to Day 15
Time of maximum observed concentration (Tmax) | Up to Day 15
Area under the concentration-time curve from time zero to time of the last quantifiable concentration (AUC(0-T)) | Up to Day 15
Total Radioactivity (TRA) | Up to Day 30

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to Day 36
Number of participants with Serious AEs (SAEs) | Up to Day 36
Number of participants with AEs leading to discontinuation | Up to Day 36
Number of participants with vital sign abnormalities | Up to Day 30
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 30
Number of participants with physical examination abnormalities | Up to Day 30
Number of participants with clinical laboratory test abnormalities | Up to Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html